CLINICAL TRIAL: NCT02602132
Title: Clamping vs. Free Drainage Before the Removal of Short-term Indwelling Urethral Catheters in Internal Medicine Patients.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants. very slow and poor recruitment
Sponsor: David Guadarrama-Ortega (Other)
Responsible Party: Sponsor-Investigator, David Guadarrama-Ortega, Registered Nurse, Hospital Universitario Fundación Alcorcón
Organization: Hospital Universitario Fundación Alcorcón (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15/63
Record Dates: First submitted 2015-11-04; First posted 2015-11-11 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Complication of Urinary Catheter
Keywords: INDWELLING URINARY CATHETER; CLAMPING; REMOVAL
MeSH Terms: interventions — Constriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clamping group (Experimental): Indwelling urinary catheter is clamped before removal and unclamped when the patient expresses his desire to urinate.
  Interventions: Procedure: Clamping
- Free drainage group (No Intervention): The urinary catheter will be removed without prior clamping.

INTERVENTIONS:
Procedure: Clamping — To clamp before the removal of short-term indwelling urethral catheters
  Arms: Clamping group

SUMMARY:
The study will be conducted at University Hospital Alcorcón Foundation, belonging to the public network of hospitals of Madrid Health Service.

The aim of this study is to evaluate the effects of clamping the urethral catheter prior to removal and determine which of the two options (clamping or free drainage) is the most recommended for removal of bladder catheterization in adults.

The interest of this study is given by the importance of proper handling of catheterization in the health of patients admitted to a hospital and are subjected to this technique. Increase its interest the need for implementation of evidence-based care, and limited scientific literature on the subject.

The study population will be patients undergoing short-term urethral catheterization at the Internal Medicine Service in the University Hospital Alcorcón Foundation.

The methodology of the study is experimental, randomized clinical trial without drug type. Interventions (prior clamped and free drainage) will be assigned in a randomized manner.

Interventions and data collection of patients who met the inclusion criteria to join the study will be conducted during 2016 and the first quarter of 2017. It is planned to present results at the end of 2017.

Keywords: BLADDER TRAINING, INDWELLING CATHETER, URINARY CATHETER, URETHRAL CATHETER, CLAMPING, REMOVAL, ACUTE URINARY RETENTION.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both sexes, aged between 18 and 85 years who require IUC 18 short-term (1 to 14 days) in the units of internal medicine at University Hospital Alcorcón Foundation.

Patients who express a desire to participate in the study by signing the informed consent.

Exclusion Criteria:

* Patients with permanent long-term (15 days or more) urinary catheter. Patients with recurrent episodes of UTI, which has submitted episodes of urinary retention in the last month, or who have urologic pathology.

Patients with cognitive impairments that hinder communication with the medical staff.

Disoriented patients in person, time and place. Anatomical and physiological genito-urinary system Alterations Patients taking a drug that affects the bladder and kidney function the week prior to catheterization.

Pregnant patients. Patients with a known history of benign prostatic hyperplasia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Incidence of recatheterization | 24h

CONTACTS AND LOCATIONS:
Overall Officials: David Guadarrama Ortega, RN, Principal Investigator — HUFA
Locations (1):
- Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid, Spain

REFERENCES:
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246